CLINICAL TRIAL: NCT04017975
Title: Optical Tissue Identification for Myocardial Architecture (OPTIMA Study)
Brief Title: Optical Tissue Identification for Myocardial Architecture
Acronym: OPTIMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aditya Kaza (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Aditya Kaza, Associate in Cardiac Surgery, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P00031701; R56HL128813 (NIH)
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Ventricular Septal Defect; Complete Atrioventricular Canal; Tetralogy of Fallot With Pulmonary Stenosis
Keywords: fiberoptic confocal microscopy; cardiac surgery
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Complete atrioventricular septal defect | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into two groups using permuted block and stratified according to type of surgical repair.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and the physician reading ECGs will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Non-imaging cohort (No Intervention): There will be no intervention for the non-imaging group. Subjects will receive standard of care for cardiac surgery.
- Imaging cohort (Experimental): Up to 5mL of 1:1000 dilute fluorescite will be applied to cardiac tissue prior to imaging with Cellvizio 100 Series System with Confocal Miniprobes. The system will be used to assist the investigator with the operative course.
  Interventions: Drug: Fluorescite; Device: Cellvizio 100 Series System with Confocal Miniprobes

INTERVENTIONS:
Drug: Fluorescite — 1 mL of Fluorescite will be diluted into 1L of saline. Up to 5mLs of the 1:1000 diluted solution will be applied topically to the cardiac tissue prior to imaging.
  Other Names: fluorescein sodium
  Arms: Imaging cohort
Device: Cellvizio 100 Series System with Confocal Miniprobes — The microscopy system will image cardiac tissue.
  Arms: Imaging cohort

SUMMARY:
The goal of this study is to test the hypothesis that fiberoptic confocal microscopy (FCM) imaging during repair of common congenital heart defects is a useful adjunct for avoidance of conduction abnormalities.

DETAILED DESCRIPTION:
This is an interventional randomized controlled study to investigate the use of fiberoptic confocal microscopy (FCM) imaging for avoidance of conduction abnormalities during repair of common congenital heart defects. Study results will be compared to a cohort of similar surgical patients following standard surgical procedures where FCM was not used. We will analyze pre-and postoperative ECGs to identify conduction abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 days to less than 18 years old
* Patients with planned surgical repair of:
* Ventricular septal defect (VSD)
* Complete atrioventricular canal (CAVC)
* Tetralogy of Fallot (ToF) with pulmonary stenosis

Exclusion Criteria:

* Prior history of adverse reaction to fluorescein sodium
* Prior history of renal failure or abnormal renal function
* Baseline PR interval > 220 msec or 98% for age
* Baseline HR > 98% for age
* Underlying genetic syndrome associated with progressive AV block or sinus node dysfunction (e.g. Holt-Oram or NKX2.5)
* Any surgical repair that requires staging or palliation
* Pregnant or lactating
* Exclusions specific to type of surgical repair
* Apical muscular VSD
* ToF with pulmonary atresia

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Rate of new conduction disorders | Immediately post-surgery
  Rate of new conduction disorders post-surgery will be determined by electrophysiologist read and compared between the two groups

SECONDARY OUTCOMES:
Change in PR interval | 1 year post-surgery
  PR interval will be compared between baseline, post-op, and 1 year follow up
Change in QTc interval | 1 year post-surgery
  QTc interval will be compared between baseline, post-op, and 1 year follow up
Change in QRS interval | Approximately 5 days post-surgery and 1 year post-surgery
  QRS interval will be compared between baseline, post-op, and 1 year follow up
Degree of heart block | 1 year post-surgery
  Degree of heart block will be assessed at post-op and 1 year follow up
Pacemaker implantation | 1 year post-surgery
  Incidence of temporary and permanent pacemaker implantation will be collected
Time to temporary pacing wire removal prior to discharge | Surgery to discharge (approximately 5 days)
  If a temporary pacing wire is placed, time to removal will be collected
Residual lesion score (RLS) at discharge | Surgery to discharge (approximately 5 days)
  RLS will be compared between groups
Need for repeat bypass | 1 day
  Need for repeat bypass for residual lesions during surgery will be collected
Adverse events | 1 year post-surgery
  Rates of adverse events will be collected and compared between the two group
Ease of use | 1 day
  Surgeon feedback regarding using the FCM system will be collected using a brief survey

CONTACTS AND LOCATIONS:
Overall Officials: Aditya K Kaza, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers.